CLINICAL TRIAL: NCT05153746
Title: Comparison of Adenoma Detection Rate Between Conventional Colonoscopy and 3D Colonoscopy: a Randomized Controlled Trial
Brief Title: Adenoma Detection Rate of 3D Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 202109112DIPB
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer
Keywords: 3D Colonoscopy; Colorectal neoplasm
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: 3D-colonoscopy vs. conventional 2D-colonoscopy Setting: Multi-centers
  Eligibility:
  Age 40 or above Indication for colonoscopy, including screening, surveillance, symptomatic, etc
  Exclusion:
  Poor and inadequate bowel preparation Incomplete study because of obstructive lesion, including cancer, stenosis, etc.
  Failure of cecal intubation, difficult insertion Inflammatory bowel disease Hereditary polyposis, (FAP, Lynch syndrome, hyperplastic polyposis, etc.)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D colonoscopy (Experimental): Colonoscopy insertion under regular method. After reaching cecum, the subjects will be randomized into 3D or conventional colonoscopy.
  Subjects in 3D colonoscopy arm:
  Colonoscopist will switch the image to 3D imaging form and wearing special glasses to enhance the 3D imaging. The 3D mode will be maintained during the whole colonoscopy withdrawal. When encountering suspicious neoplasm, the colonoscopist can use any image-enhancing technique (such as NBI or indigo carmine dye) to assist the diagnosis and use standard resection procedure (such as polypectomy) to complete lesion resection if necessary. The procedure time, withdrawal time, adenoma detection rate will be recorded during the colonoscopy. The pathology specimen will be sent for histology examination and any adverse event after colonoscopy (such as bleeding or perforation) will be recorded after routine surveillance.
  Interventions: Device: 3D colonoscopy
- Conventional colonoscopy (Active Comparator): Colonoscopy insertion under regular method. After reaching cecum, the subjects will be randomized into 3D or conventional colonoscopy.
  Subjects in conventional colonoscopy arm:
  Colonoscopist will use regular colonoscopy imaging form during the whole colonoscopy withdrawal. When encountering suspicious neoplasm, the colonoscopist can use any image-enhancing technique (such as NBI or indigo carmine dye) to assist the diagnosis and use standard resection procedure (such as polypectomy) to complete lesion resection if necessary. The procedure time, withdrawal time, adenoma detection rate will be recorded during the colonoscopy. The pathology specimen will be sent for histology examination and any adverse event after colonoscopy (such as bleeding or perforation) will be recorded after routine surveillance.
  Interventions: Device: 3D colonoscopy

INTERVENTIONS:
Device: 3D colonoscopy — 3D colonoscopy is a new device to enhance endoscopic imaging.

SUMMARY:
Adenoma detection rate (ADR) has been the most important quality indicator on colonoscopy because ADR was reversely related with CRC incidence and mortality. Several image enhanced technologies, such as narrow-band imaging (NBI) or linked colour imaging (LCI) had been proved to have ability to increase the ADR. 3D techonology, however, has not been validated on colonoscopy performance. Therefore, current study was to compare the ADR between new 3D colonoscopy and conventional 2D colonoscopy.

DETAILED DESCRIPTION:
An accumulating body of evidence has shown that detection and resection of pre-cancerous adenoma by colonoscopy could effectively prevent colorectal cancer (CRC) and its related mortality. Among various colonoscopy quality indicators, such as cecal intubation rate, withdrawal time, and adenoma detection rate (ADR), ADR is the most important one and most closely associated with the subsequent risk of CRC. A recent study further demonstrated the improvement of ADR could reduce subsequent risk of CRC.

To be noted, among all colorectal neoplasm, non-polypoid lesions, such as flat or depressed lesions, carries higher likelihood to be overlooked during conventional colonoscopy and these overlooked lesions were the main etiology of post-colonoscopy colorectal cancer (PCCRC). Nowadays, several colonoscopy technologies had been developed to enhance the detection of colorectal adenoma such as using digital or dye-spray chromoendoscopy or add-on device such as Cap-assisted endoscopy. Among them, some had showed the potential to enhance the detection of non-polypoid lesion, for example, the next-generation NBI or iSCAN.

3D endoscopy is a new technology that using image processing technique to offer more information on tissue depth in comparison with conventional 2D endoscopy. The utility of 3D endoscopy on GI tract was mainly from upper GI tract and it was proved to enhance the diagnostic accuracy on superficial gastric tumors and shortened the procedure time during performing gastric endoscopic submucosal dissection(ESD). However, few is known that whether 3D colonoscopy could enhance the adenoma detection, especially for non-polypoid lesion detection, during colonoscopy examination. Therefore, this prospective, randomized control study is aim to demonstrate the efficacy of 3D colonoscopy on adenoma detection in comparison with conventional 2D colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or above
* Indication for colonoscopy, including screening, surveillance, symptomatic, etc

Exclusion Criteria:

* Poor and inadequate bowel preparation
* Incomplete study because of obstructive lesion, including cancer, stenosis, etc.
* Failure of cecal intubation, difficult insertion
* Inflammatory bowel disease
* Hereditary polyposis, (FAP, Lynch syndrome, hyperplastic polyposis, etc.)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 1 week
  The number of subjects with at least one adenomatous polyp found during the colonoscopy

SECONDARY OUTCOMES:
Proximal adenoma detection rate | 1 weeks
  The number of subjects with at least one adenomatous polyp found at proximal colon ( cecum, ascending colon and hepatic flexure) during the colonoscopy
Sessile serrated adenoma detection rate | 1 week
  The number of subjects with at least one sessile serrated adenomatous polyp found during the colonoscopy
Adenoma per colonoscopy (APC) | 1 week
  Average adenomatous polyps number found in each colonoscopy
Flat adenoma detection rate | 1 week
  The number of subjects with at least one flat adenomatous polyp found during the colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chun Chang, AP, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan